CLINICAL TRIAL: NCT04546750
Title: Prospective Cohort Study for Varicose Veins Incidence and Natural Course
Acronym: VINCI
Status: Recruiting | Type: Observational
Sponsor: Russian Phlebological Association (Other)
Responsible Party: Sponsor
Other Study IDs: RPA 7.001.
Record Dates: First submitted 2020-09-05; First posted 2020-09-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Varicose Veins of Lower Limb; Thromboses, Venous; Venous Insufficiency
MeSH Terms: conditions — Venous Thrombosis; Venous Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without Varicose Veins: Individuals who do not have varicose veins of lower legs: C0, C1 classes according to Clinical, Etiologic, Anatomic and Pathophysiologic classification (CEAP)
- Patients with Varicose Veins: Individuals who have varicose veins of lower legs: C2 Ep class according to Clinical, Etiologic, Anatomic and Pathophysiologic classification (CEAP)

SUMMARY:
A prospective study of individuals without varicose veins and who have primary varicose veins to assess the morbidity, risk factors and natural course of chronic lower limb vein disease.

DETAILED DESCRIPTION:
Multicenter prospective cohort observational study based on a termless epidemiological registry. Periodic inspection and collection of data from the subjects is carried out annually, in the last quarter of the current year. Patient data is recorded in a digital database and is constantly updated

ELIGIBILITY:
Inclusion Criteria:

* A family members of the researcher (spouse, childrens, brothers and sisters, parents) or the researcher himself
* The possibility of annual clinical and ultrasound assessment of the venous system of the observed individuals

Exclusion Criteria:

* Any invasive treatment of the chronic venous disorder in anamnesis
* Venous thrombosis in the anamnesis or at the time of inclusion

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The main cohort is formed from those who do not have varicose veins, who are affected by different factors that we register (various physical activities, the presence or absence of pregnancy, etc.).
  An additional cohort is formed from those who have varicose veins at the time of inclusion.
  The goal is to track the natural evolution (progression) of the disease, to evaluate the incidence and risk factors of complications.
  An extremely important criterion for the formation of the study population is the possibility to control the lower legs veins of observed individuals by a qualified vascular specialist. To date, a qualitative assessment of veins according to the CEAP classification is a weak point in longitudinal epidemiological studies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary varicose veins | 1 year
  Number of Participants with the first identified varicose veins (class C2 according to CEAP classification)

SECONDARY OUTCOMES:
Progression of primary varicose veins | 1 year
  The presence of varicose veins in new areas of the lower extremites (each limb is divided into 8 areas: thigh - anterior, posterior, medial, lateral area; lower leg - anterior, posterior, medial, lateral area)
Incidence of chronic venous insufficiency | 1 year
  Number of participants with the first identified sign of chronic venous insufficiency (venous edema, venous eczema, hyperpigmentation of the skin, lipodermatosclerosis, venous ulcer)
Incidence of superficial vein thrombosis | 1 year
  Number of participants with first episode of superficial vein thrombosis
Incidence of reticular and telangiectatic leg veins | 1 year
  Number of Participants with the first identified eticular and telangiectatic leg veins ((class C1 according to CEAP classification)
Progression of reticular and telangiectatic leg veins | 1 year
  The presence of reticular and telangiectatic leg veins in new areas of the lower extremites (each limb is divided into 8 areas: thigh - anterior, posterior, medial, lateral area; lower leg - anterior, posterior, medial, lateral area)

CONTACTS AND LOCATIONS:
Locations (1):
- "Medalp" private surgery clinic, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The accumulation of data will be carried out on the basis of an termless Russian epidemiological registry, ClinicalTrials.gov Identifier: NCT04487314 — https://epid.venousregistry.org/